CLINICAL TRIAL: NCT00613834
Title: Intrauterine Lidocaine Infusion for Pain Management During Outpatient Essure Transcervical Tubal Sterilization Procedures
Brief Title: Intrauterine Lidocaine Infusion for Essure Sterilization Procedures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Alison Edelman, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: OHSU FAMPLAN 3343
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Results first posted 2019-12-19 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Pain
Keywords: Essure sterilization; pain management; intrauterine lidocaine infusion
MeSH Terms: conditions — Pain; Agnosia | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine group (Experimental): Participants receive transcervical instillation of 5 ml 4% lidocaine solution 3 minutes prior to transcervical tubal sterilization
  Interventions: Drug: Lidocaine
- Control group (Placebo Comparator): Participants receive transcervical instillation of 5 ml saline 3 minutes prior to transcervical tubal sterilization
  Interventions: Drug: Sterile Saline

INTERVENTIONS:
Drug: Lidocaine — 5 ml intrauterine infusion of 4% lidocaine using a sterile 3 mm Novak curette will be infused slowly over 4 1/2 minutes
  Other Names: Xylocaine
  Arms: Lidocaine group
Drug: Sterile Saline — 5 ml intrauterine infusion of sterile saline using a sterile 3 mm Novak curette will be infused slowly over 4 1/2 minutes
  Arms: Control group

SUMMARY:
The purpose of this study is to assess the level of pain women experience with an Essure procedure and the effect that lidocaine might have on that pain. We will also assess the absorption of lidocaine in the uterus by measuring lidocaine levels in the blood.

DETAILED DESCRIPTION:
We intend to conduct a randomized, blinded, and placebo- controlled clinical trial at Oregon Health and Science University and Planned Parenthood of the Columbia Willamette to determine if intrauterine lidocaine infusion will decrease the amount of pain subjects experience during and after Essure transcervical tubal sterilization.

We plan to enroll women who have selected Essure as their method of tubal sterilization who will be randomized to one of two groups on the days of their procedures. Subjects in Group 1, the treatment group, will receive a standard paracervical block with lidocaine intrauterine infusion and subjects in Group 2, the control group, will receive a standard paracervical block with saline intrauterine infusion. The subjects will be asked to rate their pain on a 100 mm Visual Analog Scale (VAS) at five points during the procedure and once thirty minutes following the procedure. Subjects will also be asked to rate their overall satisfaction with their care prior to leaving the recovery room.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18 or older
* Good general health, based on the opinion of the investigator
* Voluntarily requesting permanent sterilization
* Negative pregnancy test
* Agree to premedication with ibuprofen and ativan
* English speaking, or other language if an interpreter is available to be present at all points of the study procedure.
* Willing and able to sign an informed consent
* Willing to comply with the terms of the study

Exclusion Criteria:

* Significant physical or mental health condition, based on the opinion of the investigator.
* Positive pregnancy test
* Request for IV/IM sedation prior to the start of the procedure
* Refusal of ibuprofen, ativan, or paracervical block
* Allergy to any study medication including lidocaine, ibuprofen, ativan, sodium bicarbonate
* History of toxic reaction to local anesthetics
* Known hepatic disease or liver dysfunction. (Lidocaine is metabolized by the liver.)
* Weight less than 100 pounds. [Any patient weighing less than 100 pounds would receive more than the recommended dose for their weight (4.5 mg/kg or 2 mg/lb)].
* Current participation in another research study which would interfere with the conduct of this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle M. Isley, M.D., Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Planned Parenthood of the Columbia Willamette, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon

REFERENCES:
- [Derived] Isley MM, Jensen JT, Nichols MD, Lehman A, Bednarek P, Edelman A. Intrauterine lidocaine infusion for pain management during outpatient transcervical tubal sterilization: a randomized controlled trial. Contraception. 2012 Mar;85(3):275-81. doi: 10.1016/j.contraception.2011.06.015. Epub 2011 Aug 17. PMID 22067774
- See also: (Women's Health Research Unit website) — http://www.ohsuwomenshealth.com/research/index.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Saline Group: Participants receive transcervical instillation of 5 ml saline 3 minutes prior to transcervical tubal sterilization
Period: Overall Study
Arm/Group | Lidocaine Group | Saline Group
Started | 29 | 29
Completed | 29 | 26
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine Group | Saline Group | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 29 | 58
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (6.6) | 33.8 (6.3) | 33.6 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 58
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient-perceived Pain Between Baseline and Cannulization
Description: Patients rated their pain following speculum insertion (used as baseline) and after insertion of a cannula into both fallopian tubes. Reported pain during cannulization of the right and left fallopian tubes were averaged to obtain the measurement of pain at cannulization. Pain was reported using a Visual Analog Scale (VAS, range 0-100), where a score of 0 indicates no pain and a score of 100 indicates the worst pain imaginable. Baseline pain levels were subtracted from average pain during cannulization: a negative change in VAS score between baseline and cannulization indicates less pain during cannulization and a positive change in VAS score indicates more pain during cannulization.
Time Frame: Immediately after speculum insertion and immediately after cannulization
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Lidocaine Group | Saline Group
Number analyzed (Participants) | 29 | 26
score on a scale | 29.5 [-7 to 73] | 35 [-18.5 to 82]

2. Secondary Outcome: Patient Perceived Pain 30 Minutes Post-procedure
Description: Patients rated their pain 30 minutes after speculum removal using a Visual Analog Scale (VAS, range 0-100), where a score of 0 indicates no pain and a score of 100 indicates the worst pain imaginable.
Time Frame: 30 minutes post-procedure
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Lidocaine Group | Control Group
Number analyzed (Participants) | 29 | 26
score on a scale | 20 [1 to 76] | 32.5 [0 to 97]

3. Secondary Outcome: Patient Satisfaction With the Essure Tubal Sterilization Procedure
Description: Patients reported their overall satisfaction with the Essure tubal sterilization procedure using a Visual Analog scale (VAS), range 0-100. A score of 0 indicates lowest possible satisfaction and a score of 100 indicates highest possible satisfaction.
Time Frame: 30 minutes post-procedure
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Lidocaine Group | Saline Group
Number analyzed (Participants) | 29 | 29
score on a scale | 94 [46 to 100] | 93.5 [66 to 99]

ADVERSE EVENTS:
Time Frame: From enrollment to 30 minutes post-procedure
Arm/Group | Lidocaine Group | Saline Group
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29

LIMITATIONS AND CAVEATS:
Difference in reported abortions between the two groups. Data not included on three subjects in saline group because the subjects could not tolerate the procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No